CLINICAL TRIAL: NCT01838512
Title: Prospective Research Assessment in Multiple Myeloma: An Observational Evaluation (PREAMBLE)
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA204-008
Record Dates: First submitted 2013-04-19; First posted 2013-04-24 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: Participants with relapsed/refractory multiple myeloma (RRMM) followed up for up to 5 years
- Cohort 2: Participants with newly-diagnosed multiple myeloma (NDMM) followed up for up to 8 years

SUMMARY:
The purpose of this study is to assess the clinical effectiveness of all approved multiple myeloma (MM) therapies in the newly-diagnosed (NDMM) and the relapsed/refractory MM (RRMM) settings in real-world clinical practice.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

For RRMM participants who have received at least one prior line of therapy (LoT) for MM:

* Have documented progression from a prior LoT
* Participants who have initiated treatment with one of the following therapies within 90 days before consent for this study OR in the case where treatment has not yet been initiated, documentation that the treatment strategy was determined before consent for this study must be provided, and treatment must be initiated within 30 days after consent:
* IMiDs
* PIs
* Combination of IMiD + PI
* Newer agents with novel MOAs alone or in combination (eg, mAbs, HDACIs, Akt inhibitors, SINE, or CAR T-cell therapies)

For NDMM participants receiving frontline therapy:

* Eligible to receive frontline therapy for MM (no prior MM treatment)
* Participants who have initiated treatment for MM with one of the following therapies within 90 days before consent for this study OR in the case where treatment has not yet been initiated, documentation that the treatment strategy was determined before consent for this study must be provided, and treatment must be initiated within 30 days after consent:
* IMiDs
* PIs
* Combination of IMiD + PI
* Newer agents with novel MOAs alone or in combination (eg, mAbs, HDACIs, Akt inhibitors, SINE, or CAR T-cell therapies)

Exclusion Criteria:

* Participants who are currently participating in a clinical trial for MM
* Participants who are currently receiving treatment for primary cancer other than MM
* Participants who are not willing or able to provide informed consent
* Participants who are incarcerated
* Participants under compulsory detention for treatment of a physical (eg, infectious) or psychiatric illness

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of two cohorts: Participants with relapsed/refractory (RR) multiple myeloma (MM) and those with newly-diagnosed (ND) multiple myeloma (MM).
Sampling Method: Non-Probability Sample
Enrollment: 2555 (Estimated)
Dates: Start 2012-06-13 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) for participants with relapsed/refractory multiple myeloma (RRMM) | Up to 5 years
Overall Survival (OS) for participants with newly-diagnosed multiple myeloma (NDMM) | Up to 8 years
Progression-Free Survival (PFS) for participants with RRMM | Up to 5 years
Progression-Free Survival (PFS) for participants with NDMM | Up to 8 years

SECONDARY OUTCOMES:
Treatment patterns of approved MM therapies as measured by the Response Rate for participants with RRMM | From study index date until the enrollment date, assessed up to 5 years
Treatment patterns of approved MM therapies as measured by the Response Rate for participants with NDMM | From study index date until the enrollment date, assessed up to 8 years
Healthcare resource utilization (HCRU) for participants with RRMM | Up to 5 years
Healthcare resource utilization (HCRU) for participants with NDMM | Up to 8 years
Healthcare resource utilization (HCRU) for participants with RRMM | From the day of enrollment until death, withdrawal of consent, enrollment into a clinical trial for MM, loss to follow-up, or end of study, whichever comes first; assessed up to 60 months
Healthcare resource utilization (HCRU) for participants with NDMM | From the day of enrollment until death, withdrawal of consent, enrollment into a clinical trial for MM, loss to follow-up, or end of study, whichever comes first; assessed up to 96 months
Patient reported outcomes as measured by EQ-5D summary index for participants with RRMM | From start of initial therapy to questionnaire completion, assessed up to 5 years
Patient reported outcomes as measured by EQ-5D summary index for participants with NDMM | From start of initial therapy to questionnaire completion, assessed up to 8 years
Patient reported outcomes as measured by EORTC-QLQ-C30 for participants with RRMM | From start of initial therapy to questionnaire completion, assessed up to 5 years
Patient reported outcomes as measured by EORTC-QLQ-C30 for participants with NDMM | From start of initial therapy to questionnaire completion, assessed up to 8 years
Patient reported outcomes as measured by EORTC-QLQ-MY20 for participants with RRMM | From start of initial therapy to questionnaire completion, assessed up to 5 years
Patient reported outcomes as measured by EORTC-QLQ-MY20 for participants with NDMM | From start of initial therapy to questionnaire completion, assessed up to 8 years
Incidence of Adverse Events (AEs) for participants with RRMM | Up to 5 years
Incidence of Adverse Events (AEs) for participants with NDMM | Up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (125):
- United States (74):
  - Local Institution, Birmingham, Alabama
  - Local Institute, Goodyear, Arizona
  - Local Institution - 0023, Anaheim, California
  - Local Institution, Anaheim, California
  - Local Institution - 0045, Burbank, California
  - Local Institution, Corona, California
  - Local Institution - 0048, Downey, California
  - Local Institution - 0052, Fountain Valley, California
  - Local Institute, Los Angeles, California
  - Local Institute, Santa Rosa, California
  - Local Institution - 0051, Santa Rosa, California
  - Local Institution, Brooksville, Florida
  - Local Institution - 0044, Fort Lauderdale, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institute, Valdosta, Georgia
  - Local Institution - 0047, Valdosta, Georgia
  - Local Institution, Skokie, Illinois
  - Local Institution - 0041, Springfield, Illinois
  - Local Institution - 0058, Anderson, Indiana
  - Local Institution - 0011, Indianapolis, Indiana
  - Local Institution, Indianapolis, Indiana
  - Local Institute, Sioux City, Iowa
  - Local Institute, Louisville, Kentucky
  - Local Institution - 0042, Louisville, Kentucky
  - Local Institution, Lafayette, Louisiana
  - Local Institution, Shreveport, Louisiana
  - Local Institution, Minneapolis, Minnesota
  - Local Institution - 0030, Woodbury, Minnesota
  - Local Institute, Southaven, Mississippi
  - Local Institute, Kansas City, Missouri
  - Local Institution - 0050, Kansas City, Missouri
  - Local Institution - 0037, Missoula, Missouri
  - Local Institute, Saint Joseph, Missouri
  - Local Institution - 0020, Springfield, Missouri
  - Local Institution, Springfield, Missouri
  - Local Institution, St Louis, Missouri
  - Local Institute, Missoula, Montana
  - Local Institute, Omaha, Nebraska
  - Local Institution - 0024, Omaha, Nebraska
  - Local Institution - Canada, No City Provided, New Jersey
  - Local Institution - France, No City Provided, New Jersey
  - Local Institution - Germany, No City Provided, New Jersey
  - Local Institution - Italy, No City Provided, New Jersey
  - Local Institution - United Kingdom, No City Provided, New Jersey
  - Local Institution - USA, No City Provided, New Jersey
  - Local Institution - 0049, Stony Brook, New York
  - Local Institute, Cary, North Carolina
  - Local Institution - 0033, Cary, North Carolina
  - Local Institution - 0010, Gastonia, North Carolina
  - Local Institution, Gastonia, North Carolina
  - Local Institute, Canton, Ohio
  - Local Institution - 0022, Canton, Ohio
  - Local Institute, Cleveland, Ohio
  - Local Institute, Tulsa, Oklahoma
  - Local Institute, Portland, Oregon
  - Local Institute, Pottstown, Pennsylvania
  - Local Institute, Charleston, South Carolina
  - Local Institution - 0016, Charleston, South Carolina
  - Local Institute, Knoxville, Tennessee
  - Local Institution, Memphis, Tennessee
  - Local Institute, Amarillo, Texas
  - Local Institute, Corpus Christi, Texas
  - Local Institute, Dallas, Texas
  - Local Institution - 0025, Dallas, Texas
  - Local Institution - 0014, Dallas, Texas
  - Local Institution - 0032, Garland, Texas
  - Local Institute, San Antonio, Texas
  - Local Institution - 0027, San Antonio, Texas
  - Local Institute, Sherman, Texas
  - Local Institute, Seattle, Washington
  - Local Institute, Spokane, Washington
  - Local Institution - 0026, Spokane, Washington
  - Local Institute, Yakima, Washington
  - Local Institution - 0031, Yakima, Washington
- Canada (3):
  - Local Institute, Toronto, Ontario
  - Local Institution - 0066, Toronto, Ontario
  - Local Institute, Weston, Ontario
- France (8):
  - Local Institute, Blois
  - Local Institute, Chalon-sur-Saône
  - Local Institution - 0100, La Roche-sur-Yon
  - Local Institute, La Roche-sur-Yon
  - Local Institute, Limoges
  - Local Institute, Meaux
  - Local Institute, Nantes
  - Local Institute, Rennes
- Germany (11):
  - Local Institute, Heidelberg, Baden-Wurttemberg
  - Local Institute, Hamm, North Rhine-Westphalia
  - Local Institute, Aschaffenburg
  - Local Institute, Berlin
  - Local Institute, Dresden
  - Local Institution - 0070, Hamm
  - Local Institute, Magdeburg
  - Local Institution - 0067, Magdeburg
  - Local Institute, München
  - Local Institute, Rostock
  - Local Institution - 0085, Wiesbaden
- Italy (22):
  - Local Institute, Pesaro, Pesaro E Urbino
  - Local Institute, Ancona
  - Local Institution - 0119, Cagliari
  - Local Institute, Cagliari
  - Local Institution - 0111, Florence
  - Local Institute, Florence
  - Local Institute, Lecce
  - Local Institution - 0120, Messina
  - Local Institute, Milan
  - Local Institution - 0116, Milan
  - Local Institute, Napoli
  - Local Institution - 0114, Napoli
  - Local Institution - 0115, Pesaro
  - Local Institution - 0121, Pescara
  - Local Institute, Roma
  - Local Institution, Roma
  - Local Institution - 0107, Terni
  - Local Institute, Terni
  - Local Institute, Torino
  - Local Institution - 0112, Torino
  - Local Institute, Vicenza
  - Local Institution - 0117, Vicenza
- United Kingdom (7):
  - Local Institute, Truro, Cornwall
  - Local Institute, Leeds
  - Local Institution, Liverpool
  - Local Institute, Nottingham
  - Local Institution - 0095, Nottingham
  - Local Institute, Stafford
  - Local Institute, Swansea

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html